CLINICAL TRIAL: NCT04011306
Title: A Multicenter, Prospective, Randomized, Comparative Feasibility Study of a Novel Phototherapy System for the Management of Acute Burns
Brief Title: A Feasibility Study of a Novel Phototherapy System for the Management of Acute Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rogers Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP-06-001
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Burn Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lumina24 BLU (Experimental): Each subject will be randomized to receive standard of care dressing on approximately half of the study burn site, and Lumina24TM BLU treatment on the remaining half of the study burn site.
  Interventions: Device: Lumina24 BLU

INTERVENTIONS:
Device: Lumina24 BLU — Lumina24 BLU is the technology used to deliver continuous low-irradiance phototherapy for the treatment of acute burns

SUMMARY:
The primary purpose of this feasibility study is to evaluate safety and effectiveness in healing outcomes of patients treated with Lumina24TM BLU (treatment), a Continuous Low-Irradiance Phototherapy (CLIP) device, as compared to standard of care (SOC) therapy (control) for the treatment of acute burns.

DETAILED DESCRIPTION:
This feasibility study will consist of up to 15 subjects (Cohort I: up to 10 subjects with partial thickness second-degree burns; Cohort II: up to 5 subjects with deep partial thickness second- and/or full thickness third-degree burns). Each subject will be randomized to receive standard of care dressing on approximately half of the study burn site, and Lumina24TM BLU treatment on the remaining half of the study burn site. If the subject has bilaterally symmetric burns, they will be randomized to receive SOC or Lumina24TM BLU at the distinct anatomical burn locations (e.g. right/left thigh, right/left shoulder, etc.). The proposed feasibility study will inform critical primary and secondary outcome measures and procedural improvements necessary for a pivotal clinical study that would demonstrate both antimicrobial effectiveness and improved wound healing of acute burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age > 18 to < 65
* BMI > 20 kg/m2
* Patients anticipated to receive inpatient care for a minimum of 72 hours at the respective medical facility for partial thickness second-degree, deep partial thickness second-degree and/or full thickness third-degree burn wounds.
* Patients who have a > 5% to < 50% Total Body Surface Area (TBSA) wound.
* Patients are willing and able to adhere to the therapy and protocol.
* Female of childbearing potential must be willing to use acceptable methods of contraception.
* Patients may or may not have clinical signs and symptoms of burn site infection at baseline.
* Subject has read, understood and signed the approved ICF before screening procedures either by the patient or their legally authorized representative.

Exclusion Criteria:

* Subjects with burns > third-degree (i.e. involvement of deeper tissues, such as muscle, tendons, or bone)
* Patients deemed not medically stable by the treating Investigator.
* Patients with burn wounds limited to their head or genitalia.
* Patients currently enrolled or participating in another investigational device, drug or biological trial that would interfere with the Lumina24TM application.
* Patients with inhalation burns.
* Patients who are clinically septic.
* Patients are pregnant.
* Patients on a ventilator, who are undergoing acute fluid resuscitation, are hemodynamically unstable or are deemed 'comfort measures only'.
* In the opinion of treating physician, patient not expected to survive beyond 30 days.
* Pregnant or lactating status. Pregnancy as determined by a positive pregnancy test at screening or baseline.
* Known history of HIV infection, or active Hepatitis B or Hepatitis C infection.
* Cancer requiring chemotherapy or radiation within previous 6 months or resection within the last 5 years (other than basal cell carcinoma.
* Known chronic renal failure (serum creatine > 2 mg/dL) or chronic liver disease.
* Pre-existing medical condition requiring current use of immunosuppressive medication or systemic steroids
* Pre-existing medical conditions that would interfere with wound healing (i.e. diabetic patients with Hemoglobin A1c test result > 8%, malignancy, autoimmune disease)
* Subjects with psychiatric conditions that are anticipated to result in protocol noncompliance
* Chronic illicit drug or alcohol abuse that is anticipated to interfere with patient compliance with the protocol
* Subject is incarcerated at the time of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | up to 28 days
  Percentage area reduction (PAR) of the acute burn wound (SOC control site vs. Lumina24TM BLU treatment site)
Number of adverse events | up to 28 days
  Safety measured by incidence of product-related AEs, SAEs, and UADEs
Microbial load counts (Cohort II only) | up to 28 days
  Difference of bioburden in/on the burn wound (SOC control site vs. Lumina24TM BLU treatment site) assessed by quantitative analysis of microbial load counts obtained from 3-mm punch biopsies and wound cultures

SECONDARY OUTCOMES:
Time to healing | 12 months
  Time to burn wound healing at end of inpatient treatment
Numerical Pain Rating Scale | 12 months
  Difference in pain related to acute burn wounds between SOC control site and Lumina24TM BLU treatment site assessed by patient-reported rating ranging from 0 to 10 (where 0 represents no pain and 10 represents worst possible pain)
Cost-effectiveness | 12 months
  Difference in cost-effectiveness of treatment regime between Lumina24TM BLU and SOC control assessed by difference in sum of costs associated with each treatment regime (including costs of OR visits required, inpatient stay, grafts and/or biologics used)
Patient and Observer Scar Assessment Scale | 12 months
  Difference in healing of hypertrophic scarring between SOC control site and Lumina24TM BLU treatment site assessed by Patient and Observer Scar Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: David W. Mozingo, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States